CLINICAL TRIAL: NCT05493787
Title: Nudging Flu Vaccination by Making it Easy for Patients to Schedule a Flu Shot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Massachusetts Institute of Technology (Other); National Bureau of Economic Research, Inc. (Other)
Responsible Party: Principal Investigator, Christopher F Chabris, PhD, Professor, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0500
Record Dates: First submitted 2022-08-02; First posted 2022-08-09 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Influenza
Keywords: Vaccination; Health promotion; Health behavior; Economics, Behavioral
MeSH Terms: conditions — Influenza, Human; Health Behavior; Behavior

STUDY DESIGN:
Masking Description: Although patients will not be explicitly informed of which arm they were randomized to, they will be aware of the messages they receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Passive control (No Intervention): No message
- Active control message (Active Comparator): A message that simply states that patients can get a flu shot at Geisinger
  Interventions: Behavioral: Reminder
- Ease message (Experimental): A message emphasizing the ease of scheduling a flu shot at Geisinger
  Interventions: Behavioral: Reminder
- Waiting for you message (Experimental): A message that states the patient's flu shot is "waiting" for them at Geisinger
  Interventions: Behavioral: Reminder
- Protect yourself - rare message (Experimental): A message that emphasizes the rare, dangerous outcomes of getting the flu (e.g., hospitalization, pneumonia), and states that a flu shot can offer protection from those outcomes
  Interventions: Behavioral: Reminder
- Protect yourself - frequent message (Experimental): A message that emphasizes the outcomes that frequently occur in people with the flu (e.g., fever, chills, missing important events), and states that a flu shot can offer protection from those outcomes
  Interventions: Behavioral: Reminder

INTERVENTIONS:
Behavioral: Reminder — Patient portal, SMS, email, and/or another modality
  Arms: Active control message; Ease message; Protect yourself - frequent message; Protect yourself - rare message; Waiting for you message

SUMMARY:
The purpose of this study is to test whether messages that make it easy to schedule a flu shot appointment will increase flu shot rates in patients without an upcoming appointment. The study will also test which message versions and message timing are most effective for increasing flu vaccination.

DETAILED DESCRIPTION:
The CDC recommends a flu vaccination to everyone aged 6+ months, with rare exception; almost anyone can benefit from the vaccine, which can reduce illnesses, missed work, hospitalizations, and death. Past work from the study team focused on encouraging flu shots for patients with upcoming appointments. However, many patients in the health system do not have any appointments during flu season.

Eligible patients without an upcoming appointment will be randomized to a passive control group (no message), an active control group (a basic message stating that the patient can get a flu shot at Geisinger) or one of several other messages informed by behavioral science ("ease", "waiting for you", "protect yourself - rare outcomes", or "protect yourself - frequent outcomes"). Patients will be randomly assigned to one of several message send dates. Messages sent via patient portal, short message service (SMS) text, email, and/or another modality, will include a link redirecting patients to a page where they can self-schedule a flu shot.

ELIGIBILITY:
Inclusion Criteria:

* Included in one or both of the following two base patient lists:

  1. Geisinger patient portal flu outreach list for Fall 2022
  2. A list of patients obtained from Geisinger's Phenomics and Clinical Data Core (PACDC). This list will include active Geisinger patients (all patients on this list attended at least one primary care appointment at Geisinger between 10/1/2008 and 4/13/2022, and either had a Geisinger primary care provider assigned as of April 2022, or were in the Electronic Health Record [EHR] since at least September 2021 and had at least one encounter in 2020-2022).
* Aged 18 or older as of October 2022
* Has had a Geisinger encounter in the last 2 years as of October 2022
* Either of the following, as of October 2022:

  1. Has a Geisinger PCP assigned in the Community Medicine, Pediatrics, or Internal Medicine service line
  2. In the last 2 years, has completed an appointment in a Geisinger specialty on a list of specialties approved by system leadership for flu shot communications
* Has not received a flu-shot during the 2022-23 flu season as of ~1 week prior to the message date (timeline may be slightly different, depending on data pull logistics), according to the Electronic Health Record (EHR)
* Does not have a scheduled in-person primary care or in-person flu-shot-eligible specialty appointment in the 12 weeks following their assigned message send date, as of ~1 week prior to the message date (timelines may be slightly different, depending on data pull logistics or clinical guidance)

  * As of this writing, the team plans to define a flu-shot-eligible specialty appointments as appointments in departments that have historically documented or administered flu vaccine. However, this approach may change slightly based on changing clinical guidance.

Exclusion Criteria:

* The CMSL/Marketing list will include patients in Geisinger's 65Forward or Community Care populations. If necessary due to logistical constraints, we may exclude these 65Forward and/or Community Care patients from our study.
* Cannot be contacted via the communication modality being used in the study (e.g., patient portal, SMS), e.g., due to insufficient/missing contact information in the EHR or because they opted out
* Has an allergy to flu vaccines according to any EHR allergy table known to the study team
* Has a health maintenance modifier indicating they are permanently discontinued from receiving a seasonal flu shot
* Is on a list of dismissed patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139503 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher F Chabris, PhD, Principal Investigator — Geisinger Clinic; Michelle N Meyer, PhD JD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Clinic, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: By the paper's online publication date. Data will remain available for as long as the Open Science Framework hosts it.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: https://osf.io/qsemk/

RESULTS

PARTICIPANT FLOW:
Groups:
- Passive Control - November; Passive Control - December: No message
- Active Control Message - November; Active Control Message - December: A message that simply states that patients can get a flu shot at Geisinger
  Reminder: Patient portal, SMS, email, and/or another modality
- Ease Message - November; Ease Message - December: A message emphasizing the ease of scheduling a flu shot at Geisinger
  Reminder: Patient portal, SMS, email, and/or another modality
- Waiting for You Message - November; Waiting for You Message - December: A message that states the patient's flu shot is "waiting" for them at Geisinger
  Reminder: Patient portal, SMS, email, and/or another modality
- Protect Yourself - Rare Message - November; Protect Yourself - Rare Message - December: A message that emphasizes the rare, dangerous outcomes of getting the flu (e.g., hospitalization, pneumonia), and states that a flu shot can offer protection from those outcomes
  Reminder: Patient portal, SMS, email, and/or another modality
- Protect Yourself - Frequent Message - November; Protect Yourself - Frequent Message - December: A message that emphasizes the outcomes that frequently occur in people with the flu (e.g., fever, chills, missing important events), and states that a flu shot can offer protection from those outcomes
  Reminder: Patient portal, SMS, email, and/or another modality
Period: Overall Study
Arm/Group | Passive Control - November | Active Control Message - November | Ease Message - November | Waiting for You Message - November | Protect Yourself - Rare Message - November | Protect Yourself - Frequent Message - November | Passive Control - December | Active Control Message - December | Ease Message - December | Waiting for You Message - December | Protect Yourself - Rare Message - December | Protect Yourself - Frequent Message - December
Started | 12531 | 12531 | 12531 | 12531 | 12530 | 12531 | 10705 | 10743 | 10657 | 10783 | 10702 | 10728
Completed | 12531 | 12531 | 12531 | 12531 | 12530 | 12531 | 10705 | 10743 | 10657 | 10783 | 10702 | 10728
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Passive Control - November | Active Control Message - November | Ease Message - November | Waiting for You Message - November | Protect Yourself - Rare Message - November | Protect Yourself - Frequent Message - November | Passive Control - December | Active Control Message - December | Ease Message - December | Waiting for You Message - December | Protect Yourself - Rare Message - December | Protect Yourself - Frequent Message - December | Total
Number analyzed (Participants) | 12531 | 12531 | 12531 | 12531 | 12530 | 12531 | 10705 | 10743 | 10657 | 10783 | 10702 | 10728 | 139503
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 11105 | 11041 | 11096 | 11073 | 11018 | 11040 | 9573 | 9585 | 9564 | 9621 | 9532 | 9564 | 123812
  65+ years | 1426 | 1490 | 1435 | 1458 | 1512 | 1491 | 1132 | 1158 | 1093 | 1162 | 1170 | 1164 | 15691
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7019 | 7025 | 7048 | 7126 | 7047 | 7153 | 6002 | 5964 | 5945 | 6007 | 5960 | 6072 | 78368
  Male | 5512 | 5506 | 5483 | 5405 | 5483 | 5378 | 4703 | 4779 | 4712 | 4776 | 4742 | 4656 | 61135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 551 | 581 | 632 | 613 | 590 | 612 | 501 | 513 | 537 | 537 | 528 | 494 | 6689
  Not Hispanic or Latino | 11851 | 11810 | 11759 | 11783 | 11794 | 11784 | 10078 | 10119 | 10000 | 10127 | 10060 | 10126 | 131291
  Unknown or Not Reported | 129 | 140 | 140 | 135 | 146 | 135 | 126 | 111 | 120 | 119 | 114 | 108 | 1523
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 21 | 20 | 29 | 41 | 27 | 35 | 25 | 30 | 19 | 33 | 20 | 22 | 322
  Asian | 159 | 195 | 183 | 181 | 154 | 173 | 128 | 145 | 131 | 139 | 157 | 146 | 1891
  Native Hawaiian or Other Pacific Islander | 50 | 56 | 57 | 64 | 50 | 48 | 52 | 62 | 51 | 46 | 37 | 54 | 627
  Black or African American | 508 | 505 | 542 | 507 | 484 | 534 | 460 | 444 | 466 | 450 | 451 | 422 | 5773
  White | 11636 | 11604 | 11575 | 11566 | 11646 | 11592 | 9914 | 9937 | 9857 | 9980 | 9880 | 9962 | 129149
  More than one race | 4 | 5 | 3 | 4 | 1 | 1 | 3 | 0 | 2 | 0 | 0 | 1 | 24
  Unknown or Not Reported | 153 | 146 | 142 | 168 | 168 | 148 | 123 | 125 | 131 | 135 | 157 | 121 | 1717
Region of Enrollment [Number; unit: participants]
  United States | 12531 | 12531 | 12531 | 12531 | 12530 | 12531 | 10705 | 10743 | 10657 | 10783 | 10702 | 10728 | 139503

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Self-scheduled a Flu Shot
Description: Patient self-schedules a flu vaccine appointment through the patient portal.
  This outcome measures whether the patient schedules an appointment within 4 weeks of the send date, but the appointment can occur more than 4 weeks past the send date.
Time Frame: Within 4 weeks of message send date
Measure: Count of Participants; unit: Participants
Arm/Group | Passive Control - November | Active Control Message - November | Ease Message - November | Waiting for You Message - November | Protect Yourself - Rare Message | Protect Yourself - Frequent Message - November | Passive Control - December | Active Control Message - December | Ease Message - December | Waiting for You Message - December | Protect Yourself - Rare Message - December | Protect Yourself - Frequent Message - December
Number analyzed (Participants) | 12531 | 12531 | 12531 | 12531 | 12530 | 12531 | 10705 | 10743 | 10657 | 10783 | 10702 | 10728
Participants | 43 | 63 | 62 | 74 | 70 | 53 | 8 | 28 | 36 | 44 | 20 | 26
Statistical Analysis 1: Comparison: Passive Control - November vs Active Control Message - November vs Passive Control - December vs Active Control Message - December; Null hypothesis: Flu shot self-scheduling does not differ between those sent an Active Control message and those not sent a message (i.e., those in the Passive Control group); Alternative hypothesis: Sending an Active Control message increases self-scheduling compared with sending no message. Analysis combines across November and December send dates; Test type: Superiority; p = .003, Regression, Linear — Comparisons between Passive Control and all other arms (Analyses 1-5) were analyzed in the same regression. The p-value reported is 2-tailed
Statistical Analysis 2: Comparison: Passive Control - November vs Ease Message - November vs Passive Control - December vs Ease Message - December; Null hypothesis: Flu shot self-scheduling does not differ between those sent an Ease message and those not sent a message (i.e., those in the Passive Control group); Alternative hypothesis: Sending an Ease message increases self-scheduling compared with sending no message. Analysis combines across November and December send dates; Test type: Superiority; p < .001, Regression, Linear — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Passive Control - November vs Waiting for You Message - November vs Passive Control - December vs Waiting for You Message - December; Null hypothesis: Flu shot self-scheduling does not differ between those sent an Waiting for You message message and those not sent a message (i.e., those in the Passive Control group); Alternative hypothesis: Sending a Waiting for You message increases self-scheduling compared with sending no message. Analysis combines across November and December send dates; Test type: Superiority; p < .001, Regression, Linear — Comparisons between Passive Control and all other arms (Analyses 1-5) were analyzed in the same regression
Statistical Analysis 4: Comparison: Passive Control - November vs Protect Yourself - Rare Message vs Passive Control - December vs Protect Yourself - Rare Message - December; Null hypothesis: Flu shot self-scheduling does not differ between those sent a Protect Yourself - Rare message and those not sent a message (i.e., those in the Passive Control group); Alternative hypothesis: Sending a Protect Yourself - Rare Message increases self-scheduling compared with sending no message. Analysis combines across November and December send dates; Test type: Superiority; p = .003, Regression, Linear — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Passive Control - November vs Protect Yourself - Frequent Message - November vs Passive Control - December vs Protect Yourself - Frequent Message - December; Null hypothesis: Flu shot self-scheduling does not differ between those sent a Protect Yourself - Frequent message and those not sent a message (i.e., those in the Passive Control group); Alternative hypothesis: Sending a Protect Yourself - Frequent message increases self-scheduling compared with sending no message. Analysis combines across November and December send dates; Test type: Superiority; p = .035, Regression, Linear — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Active Control Message - November vs Ease Message - November vs Active Control Message - December vs Ease Message - December; Null hypothesis: Active Control messages and Ease messages are equally effective at promoting flu shot self-scheduling; Alternative hypothesis: Ease messages are more effective at promoting flu shot self-scheduling than Active Control messages. Analysis combines across November and December send dates; Test type: Superiority; p = .593, Regression, Linear — Comparisons between Active Control and all other arms (Analyses 6-9) were analyzed in the same regression. The p-value reported is 2-tailed
Statistical Analysis 7: Comparison: Active Control Message - November vs Waiting for You Message - November vs Active Control Message - December vs Waiting for You Message - December; Null hypothesis: Active Control messages and Waiting for You messages are equally effective at promoting flu shot self-scheduling; Alternative hypothesis: Waiting for You messages are more effective at promoting flu shot self-scheduling than Active Control messages. Analysis combines across November and December send dates; Test type: Superiority; p = .052, Regression, Linear — [p-value comment as in outcome 1, analysis 6]
Statistical Analysis 8: Comparison: Active Control Message - November vs Protect Yourself - Rare Message vs Active Control Message - December vs Protect Yourself - Rare Message - December; Null hypothesis: Active Control messages and Protect Yourself - Rare messages are equally effective at promoting flu shot self-scheduling; Alternative hypothesis: Protect Yourself - Rare messages are more effective at promoting flu shot self-scheduling than Active Control messages. Analysis combines across November and December send dates; Test type: Superiority; p = .952, Regression, Linear — [p-value comment as in outcome 1, analysis 6]
Statistical Analysis 9: Comparison: Active Control Message - November vs Protect Yourself - Frequent Message - November vs Active Control Message - December vs Protect Yourself - Frequent Message - December; Null hypothesis: Active Control messages and Protect Yourself - Frequent messages are equally effective at promoting flu shot self-scheduling; Alternative hypothesis: Protect Yourself - Frequent messages are more effective at promoting flu shot self-scheduling than Active Control messages. Analysis combines across November and December send dates; Test type: Superiority; p = .386, Regression, Linear — [p-value comment as in outcome 1, analysis 6]
Statistical Analysis 10: Comparison: Ease Message - November vs Waiting for You Message - November vs Ease Message - December vs Waiting for You Message - December; Null hypothesis: Ease messages and Waiting for You messages are equally effective at promoting flu shot self-scheduling; Alternative hypothesis: There is a difference in effectiveness between Ease and Waiting for You messages. Analysis combines across November and December send dates; Test type: Superiority; p = .498, Regression, Linear — Pairwise comparisons between experimental arms (Analyses 10-15) were analyzed in the same regression. Reported p-values were 2-tailed and adjusted using Tukey's HSD test
Statistical Analysis 11: Comparison: Ease Message - November vs Protect Yourself - Rare Message vs Ease Message - December vs Protect Yourself - Rare Message - December; Null hypothesis: Ease messages and Protect Yourself - Rare messages are equally effective at promoting flu shot self-scheduling; Alternative hypothesis: There is a difference in effectiveness between Ease and Protect Yourself - Rare messages. Analysis combines across November and December send dates; Test type: Superiority; p = .935, Regression, Linear — [p-value comment as in outcome 1, analysis 10]
Statistical Analysis 12: Comparison: Ease Message - November vs Protect Yourself - Frequent Message - November vs Ease Message - December vs Protect Yourself - Frequent Message - December; Null hypothesis: Ease messages and Protect Yourself - Frequent messages are equally effective at promoting flu shot self-scheduling; Alternative hypothesis: There is a difference in effectiveness between Ease and Protect Yourself - Frequent message messages. Analysis combines across November and December send dates; Test type: Superiority; p = .504, Regression, Linear — [p-value comment as in outcome 1, analysis 10]
Statistical Analysis 13: Comparison: Waiting for You Message - November vs Protect Yourself - Rare Message vs Waiting for You Message - December vs Protect Yourself - Rare Message - December; Null hypothesis: Protect Yourself - Rare and Waiting for You messages are equally effective at promoting flu shot self-scheduling; Alternative hypothesis: There is a difference in effectiveness between Protect Yourself - Rare and Waiting for You messages. Analysis combines across November and December send dates; Test type: Superiority; p = .190, Regression, Linear — [p-value comment as in outcome 1, analysis 10]
Statistical Analysis 14: Comparison: Waiting for You Message - November vs Protect Yourself - Frequent Message - November vs Waiting for You Message - December vs Protect Yourself - Frequent Message - December; Null hypothesis: Protect Yourself - Frequent messages and Waiting for You messages are equally effective at promoting flu shot self-scheduling; Alternative hypothesis: There is a difference in effectiveness between Protect Yourself - Frequent and Waiting for You messages. Analysis combines across November and December send dates; Test type: Superiority; p = .027, Regression, Linear — [p-value comment as in outcome 1, analysis 10]
Statistical Analysis 15: Comparison: Protect Yourself - Rare Message vs Protect Yourself - Frequent Message - November vs Protect Yourself - Rare Message - December vs Protect Yourself - Frequent Message - December; Null hypothesis: Protect Yourself - Rare and Protect Yourself - Frequent messages are equally effective at promoting flu shot self-scheduling; Alternative hypothesis: There is a difference in effectiveness between Protect Yourself - Rare and Protect Yourself - Frequent messages. Analysis combines across November and December send dates; Test type: Superiority; p = .854, Regression, Linear — [p-value comment as in outcome 1, analysis 10]
Statistical Analysis 16: Comparison: Passive Control - November vs Active Control Message - November vs Ease Message - November vs Waiting for You Message - November vs Protect Yourself - Rare Message vs Protect Yourself - Frequent Message - November vs Passive Control - December vs Active Control Message - December vs Ease Message - December vs Waiting for You Message - December vs Protect Yourself - Rare Message - December vs Protect Yourself - Frequent Message - December; Null Hypothesis: Messages sent in November and December are equally effective at promoting flu-shot self-scheduling. Alternative hypothesis: Messages sent in November and December are differentially effective. To test the alternative hypothesis, all message arms (Active control, Ease, Waiting for you, Protect yourself - rare, Protect yourself - frequent) were combined and compared with Passive control; Test type: Superiority; p = .637, Regression, Linear — The reported p-value (2-tailed) is for the interaction term between message send date (November, December) and message (any message arm no message)

2. Secondary Outcome: Flu Vaccination
Description: Number of patients who received a flu vaccine
Time Frame: Within 4 weeks of message send date
Measure: Count of Participants; unit: Participants
Arm/Group | Passive Control - November | Active Control Message - November | Ease Message - November | Waiting for You Message - November | Protect Yourself - Rare Message - November | Protect Yourself - Frequent Message - November | Passive Control - December | Active Control Message - December | Ease Message - December | Waiting for You Message - December | Protect Yourself - Rare Message - December | Protect Yourself - Frequent Message - December
Number analyzed (Participants) | 12531 | 12531 | 12531 | 12531 | 12530 | 12531 | 10705 | 10743 | 10657 | 10783 | 10702 | 10728
Participants | 488 | 450 | 468 | 460 | 450 | 478 | 146 | 158 | 153 | 177 | 142 | 124

3. Other Pre Specified Outcome: High Confidence Flu Diagnosis
Description: Patient received a flu diagnosis via a positive PCR/antigen/molecular test (yes/no) during the 2022-23 flu season (from the patient's message send date through April 30, 2023).
Time Frame: Up to 7 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: "Likely Flu" Diagnosis
Description: Received a "high confidence flu" diagnosis (with positive polymerase chain reaction [PCR]/antigen/molecular test) and/or "likely flu" diagnosis (as assessed via International Classification of Disease [ICD] codes or Tamiflu administration or positive PCR/antigen/molecular test) (yes/no) during the 2022-23 flu season (from the patient's message send date through April 30, 2023).
  Note that "likely flu" is a superset of the "high confidence flu" diagnoses.
Time Frame: Up to 7 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Flu Complications
Description: Diagnosed with flu-related complications (yes/no) from the patient's message send date through July 31, 2023.
Time Frame: Up to 10 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: ER Visits
Description: Number of ER visits from the patient's message send date through July 31, 2023.
Time Frame: Up to 10 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Hospitalizations
Description: Number of hospitalizations from the patient's message send date through July 31, 2023.
Time Frame: Up to 10 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: COVID-19 Vaccination Rates
Description: Received at least one COVID-19 vaccination (yes/no) during the 2022-23 flu season (from the patient's message send date through April 30, 2023).
Time Frame: Up to 7 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Number of Patients Who Self-Scheduled a Flu Shot by Sex
Description: Patient self-schedules a flu vaccine through the patient portal This outcome measures whether the patient schedules an appointment within 4 weeks of the message send date, but the appointment can occur more than 4 weeks past the send date.
Time Frame: Within 4 weeks of the message send date
Population: This outcome divides the population by sex (as listed in the electronic health record)
Measure: Count of Participants; unit: Participants
Arm/Group | Passive Control - November | Active Control Message - November | Ease Message - November | Waiting for You Message - November | Protect Yourself - Rare Message - November | Protect Yourself - Frequent Message - November | Passive Control - December | Active Control Message - December | Ease Message - December | Waiting for You Message - December | Protect Yourself - Rare Message - December | Protect Yourself - Frequent Message - December
Number analyzed (Participants) | 12531 | 12531 | 12531 | 12531 | 12530 | 12531 | 10705 | 10743 | 10657 | 10783 | 10702 | 10728
Participants
  Female: number analyzed (Participants) | 7019 | 7025 | 7048 | 7126 | 7047 | 7153 | 6002 | 5964 | 5945 | 6007 | 5960 | 6072
  Female | 28 | 38 | 46 | 45 | 53 | 31 | 6 | 13 | 21 | 25 | 11 | 9
  Male: number analyzed (Participants) | 5512 | 5506 | 5483 | 5405 | 5483 | 5378 | 4703 | 4779 | 4712 | 4776 | 4742 | 4656
  Male | 15 | 25 | 16 | 29 | 17 | 22 | 2 | 15 | 15 | 19 | 9 | 17

10. Other Pre Specified Outcome: Number of Patients Who Self-Scheduled a Flu Shot by Race
Description: as for outcome 9
Time Frame: Within 4 weeks of the message send date
Population: This outcome divides the population by race (as listed in the electronic health record)
Measure: Count of Participants; unit: Participants
Arm/Group | Passive Control - November | Active Control Message - November | Ease Message - November | Waiting for You Message - November | Protect Yourself - Rare Message - November | Protect Yourself - Frequent Message - November | Passive Control - December | Active Control Message - December | Ease Message - December | Waiting for You Message - December | Protect Yourself - Rare Message - December | Protect Yourself - Frequent Message - December
Number analyzed (Participants) | 12531 | 12531 | 12531 | 12531 | 12530 | 12531 | 10705 | 10743 | 10657 | 10783 | 10702 | 10728
Participants
  American Indian or Alaska Native: number analyzed (Participants) | 21 | 20 | 29 | 41 | 27 | 35 | 25 | 30 | 19 | 33 | 20 | 22
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian: number analyzed (Participants) | 159 | 195 | 183 | 181 | 154 | 173 | 128 | 145 | 131 | 139 | 157 | 146
  Asian | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 50 | 56 | 57 | 64 | 50 | 48 | 52 | 62 | 51 | 46 | 37 | 54
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American: number analyzed (Participants) | 508 | 505 | 542 | 507 | 484 | 534 | 460 | 444 | 466 | 450 | 451 | 422
  Black or African American | 1 | 4 | 4 | 1 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 1
  White: number analyzed (Participants) | 11636 | 11604 | 11575 | 11566 | 11646 | 11592 | 9914 | 9937 | 9857 | 9980 | 9880 | 9962
  White | 40 | 57 | 57 | 71 | 67 | 50 | 7 | 24 | 34 | 40 | 18 | 25
  Two or More: number analyzed (Participants) | 4 | 5 | 3 | 4 | 1 | 1 | 3 | 0 | 2 | 0 | 0 | 1
  Two or More | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown: number analyzed (Participants) | 153 | 146 | 142 | 168 | 168 | 148 | 123 | 125 | 131 | 135 | 157 | 121
  Unknown | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 3 | 1 | 0 | 1 | 0

11. Other Pre Specified Outcome: Number of Patients Who Self-Scheduled a Flu Shot by Ethnicity
Description: as for outcome 9
Time Frame: Within 4 weeks of the message send date
Population: This outcome divides the population by ethnicity (as listed in the electronic health record)
Measure: Count of Participants; unit: Participants
Arm/Group | Passive Control - November | Active Control Message - November | Ease Message - November | Waiting for You Message - November | Protect Yourself - Rare Message - November | Protect Yourself - Frequent Message - November | Passive Control - December | Active Control Message - December | Ease Message - December | Waiting for You Message - December | Protect Yourself - Rare Message - December | Protect Yourself - Frequent Message - December
Number analyzed (Participants) | 12531 | 12531 | 12531 | 12531 | 12530 | 12531 | 10705 | 10743 | 10657 | 10783 | 10702 | 10728
Participants
  Hispanic or Latino: number analyzed (Participants) | 551 | 581 | 632 | 613 | 590 | 612 | 501 | 513 | 537 | 537 | 528 | 494
  Hispanic or Latino | 3 | 2 | 3 | 5 | 0 | 1 | 3 | 1 | 0 | 2 | 1 | 2
  Not Hispanic or Latino: number analyzed (Participants) | 11851 | 11810 | 11759 | 11783 | 11794 | 11784 | 10078 | 10119 | 10000 | 10127 | 10060 | 10126
  Not Hispanic or Latino | 40 | 61 | 59 | 69 | 69 | 51 | 5 | 25 | 36 | 41 | 19 | 24
  Unable to Obtain: number analyzed (Participants) | 129 | 140 | 140 | 135 | 146 | 135 | 126 | 111 | 120 | 119 | 114 | 108
  Unable to Obtain | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored. See description.
Description: This is a minimal risk study, and has received expedited IRB review in keeping with 45 CFR § 46.110. EHR and claims data will report inputs (i.e., the subject's assigned arm) and outcomes (i.e., flu vaccination, flu diagnosis, flu-like symptoms). We therefore did not monitor the data for AE/SAEs.
Arm/Group | Passive Control - November | Active Control Message - November | Ease Message - November | Waiting for You Message - November | Protect Yourself - Rare Message - November | Protect Yourself - Frequent Message - November | Passive Control - December | Active Control Message - December | Ease Message - December | Waiting for You Message - December | Protect Yourself - Rare Message - December | Protect Yourself - Frequent Message - December
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-09-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT05493787/Prot_001.pdf
  • Statistical Analysis Plan (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT05493787/SAP_000.pdf